CLINICAL TRIAL: NCT01007799
Title: A Randomized, Clinical Trial of a Novel Immunotherapy for Chronic Sinusitis: Vitamin D
Brief Title: Vitamin D for Chronic Sinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16601A
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Sinusitis
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo pills to take for 12 weeks
  Interventions: Dietary Supplement: vitamin D placebo
- Vitamin D (Active Comparator): Vitamin D supplement for 12 weeks
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D placebo — 12 weeks of placebo
  Arms: Placebo
Dietary Supplement: Vitamin D — 12 weeks supplementation based on serum vitamin D levels
  Arms: Vitamin D

SUMMARY:
The purpose of this study is to examine if vitamin D improves the symptoms of chronic sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* African American (4 grandparents with AA ancestry)
* Age>18 years
* Diagnosis of chronic sinusitis

Exclusion Criteria:

* Women of childbearing potential not utilizing contraception
* Subjects with contraindications to vitamin D therapy
* History of nephrolithiasis, hypercalcemia, sarcoidosis, recent (3 month) hospitalization
* Use of immunosuppressants/medications that interfere with vitamin D metabolism (e.g., phenytoin and carbamazepine)
* Malignancy
* Kidney, gastrointestinal, or liver disorders
* Immunodeficiency
* Morbid obesity (BMI>35 kg/m2)
* Changes to medications for 6 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
score on the Sinonasal Outcome Test-22 (SNOT-22) | study onset, mid-point and conclusion

SECONDARY OUTCOMES:
Quality of life as measured by SF-36 | At entry and at completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Pinto, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States